CLINICAL TRIAL: NCT05346211
Title: The Effect of Curcumin Supplementation on Recovery From Exercise-induced Muscle Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ASE22HELCON
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Exercise Induced Muscle Damage
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Curcumin Single (Experimental): The Single dose group will consume 1 placebo sachet and one curcumin sachet per day.
  Curcumin supplementation will be from YourZooki, the supplement in question is commercially offered to the public in a tangerine flavour. The sachets will be in 750mg hydrolysed format.
  The placebo is a sachet containing the same ingredients mentioned above minus the curcumin. The sachets will be in 750mg hydrolysed format.
  Supplementation will be administered and commence 48-hours prior to the first testing day and will be consumed twice a day (8am & 8pm).
  Interventions: Dietary Supplement: Curcumin
- Curcumin Double (Experimental): The double dose group will consume two sachets per day of curcumin.
  Curcumin supplementation will be from YourZooki, the supplement in question is commercially offered to the public in a tangerine flavour. The sachets will be in 750mg hydrolysed format.
  Supplementation will be administered and commence 48-hours prior to the first testing day and will be consumed twice a day (8am & 8pm).
  Interventions: Dietary Supplement: Curcumin
- Placebo (No Intervention): Placebo sachets containing the same ingredients mentioned above minus the curcumin. The sachets will be in 750mg hydrolysed format.
  Participants will consume two sachets per day.
  Supplementation will be administered and commence 48-hours prior to the first testing day and will be consumed twice a day (8am & 8pm).

INTERVENTIONS:
Dietary Supplement: Curcumin — Curcumin Supplementation
  Arms: Curcumin Double; Curcumin Single

SUMMARY:
Recent evidence suggests that curcumin supplementation may reduce muscle inflammation, oxidative markers, and muscle damage. The most favourable dosage to elicit these ergogenic effects are yet to be established; both 750mg & 1500mg has been shown to be effective. Curcumin supplementation has been ingested in numerous different ways however, no previous research to date has used curcumin in a hydrolysed (drinkable) format. The aim of this study is to investigate whether hydrolysed curcumin can reduce indices of muscle damage and improve recovery, whilst also examining a potential dose-response effect.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are as follows:

* between the age of 18-35
* non-smoker
* no previous history of cardiovascular, respiratory, or neurological problems
* not taking anticoagulant medication
* injury-free in the 3 months prior to scheduled participation in the study

Exclusion Criteria:

Exclusion criteria include:

* hypertension (<140/80)
* any blood diseases or clotting issues,
* injury, or previous injury in <3 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood markers | Baseline
  Blood samples will be taken for analysis of markers of IL-6, IL-1β, TNF-α, IL-1, IL-4, IL-10 and CK will be taken
Blood markers | immediately post muscle damage intervention
  Blood samples will be taken for analysis of markers of IL-6, IL-1β, TNF-α, IL-1, IL-4, IL-10 and CK will be taken
Blood markers | 24 hours post
  Blood samples will be taken for analysis of markers of IL-6, IL-1β, TNF-α, IL-1, IL-4, IL-10 and CK will be taken
Blood markers | 48 hours post
  Blood samples will be taken for analysis of markers of IL-6, IL-1β, TNF-α, IL-1, IL-4, IL-10 and CK will be taken
Blood markers | 72 hours post
  Blood samples will be taken for analysis of markers of IL-6, IL-1β, TNF-α, IL-1, IL-4, IL-10 and CK will be taken
Ford and Fort | Baseline
  Capillary sample Ford and Fort tests
Ford and Fort | Immediately post muscle damage intervention
  Capillary sample Ford and Fort tests
Ford and Fort | 24 hours post
  Capillary sample Ford and Fort tests
Ford and Fort | 48 hours post
  Capillary sample Ford and Fort tests
Ford and Fort | 72 hours post
  Capillary sample Ford and Fort tests
Soreness | Baseline
  Perceived muscle soreness scale - Visual analouge scale
Soreness | Immediately post muscle damage intervention
  Perceived muscle soreness scale - Visual analouge scale
Soreness | 24 hours post
  Perceived muscle soreness scale - Visual analouge scale
Soreness | 48 hours post
  Perceived muscle soreness scale - Visual analouge scale
Soreness | 72 hours post
  Perceived muscle soreness scale - Visual analouge scale
Soreness | Baseline
  BORG CR-10 scale
Soreness | Immediately post muscle damage intervention
  BORG CR-10 scale
Soreness | 24 hours post
  BORG CR-10 scale
Soreness | 48 hours post
  BORG CR-10 scale
Soreness | 72 hours post
  BORG CR-10 scale
Soreness | Baseline
  Pressure pain threshold
Soreness | Immediately post muscle damage intervention
  Pressure pain threshold
Soreness | 24 hours post
  Pressure pain threshold
Soreness | 48 hours post
  Pressure pain threshold
Soreness | 72 hours post
  Pressure pain threshold
Muscle Structure | Baseline
  Muscle swelling - thigh girth + Ultrasound measurement
Muscle Structure | Immediately post muscle damage intervention
  Muscle swelling - thigh girth + Ultrasound measurement
Muscle Structure | 24 hours post
  Muscle swelling - thigh girth + Ultrasound measurement
Muscle Structure | 48 hours post
  Muscle swelling - thigh girth + Ultrasound measurement
Muscle Structure | 72 hours post
  Muscle swelling - thigh girth + Ultrasound measurement
Muscle Function | Baseline
  maximal strength
Muscle Function | Immediately post muscle damage intervention
  maximal strength
Muscle Function | 24 hours post
  maximal strength
Muscle Function | 48 hours post
  maximal strength
Muscle Function | 72 hours post
  maximal strength
Muscle Function | Baseline
  Muscular endurance
Muscle Function | Immediately post muscle damage intervention
  Muscular endurance
Muscle Function | 24 hours post
  Muscular endurance
Muscle Function | 48 hours post
  Muscular endurance
Muscle Function | 72 hours post
  Muscular endurance

CONTACTS AND LOCATIONS:
Overall Officials: Luke Hughes, PhD, Principal Investigator — Northumbria University; Jess Hill, PhD, Principal Investigator — St. Mary's University, Twickenham

IPD SHARING:
Plan to Share IPD: No